CLINICAL TRIAL: NCT02934958
Title: FIT Mailing Protocol-For Cancer Screening Navigation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Renown Regional Medical Center (Other)
Responsible Party: Principal Investigator, John F. Gray MD FACG AGAF, Principal Investigator, Renown Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GI-0002-1
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Neoplasms
Keywords: Colon Cancer Screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FIT Positive (Active Comparator): Referral to GI or Primary Care. Patients will be referred to MD for pre-colonoscopy vist.Standard of Care.
  Interventions: Behavioral: Standard of Care
- FIT Positive Choice (Experimental): Offered Chioce of Direct referral. Patients will be given a choice to advance to directly having a colonoscopy screening.Colon Cancer Screening Navigation.
  Interventions: Behavioral: Colon Cancer Screening Navigation

INTERVENTIONS:
Behavioral: Colon Cancer Screening Navigation — Patients with FIT Positive results that have been given the choice will be followed and navigated from referral to colonoscopy to assist in obtaining colonoscopy.
  Arms: FIT Positive Choice
Behavioral: Standard of Care — Patients will be tracked to compare how effective are usual care methods
  Arms: FIT Positive

SUMMARY:
We plan to study whether the impact of offering the choice of a pre-colonoscopy physician visit or direct referral to colonoscopy will increase adherence to colonoscopy relative to usual care in a large fecal immunochemical test (FIT) mailing campaign.

We will evaluate two study options, usual care during which patients will be required to have an office visit with wither a PCP or a Gastroenterologist prior to being scheduled for a colonoscopy, or a choice where patients will be given the option of a pre-colonoscopy visit with a gastroenterologist or PCP vs. direct referral for a colonoscopy.

In these two options we will examine colonoscopy adherence, adequacy of triage, patient satisfaction, colonoscopy outcomes (no show rate, prep quality, and pain during colonoscopy) and how insurance coverage, gender, race, education or patient understanding of colon cancer screening message during the navigation process might impact outcomes.

DETAILED DESCRIPTION:
A total of 13,392 patients will be invited to participate in the study. Approximately 2500 patients will be enrolled in the study every month for 4 months. This sampling plan will enable sufficient statistical power (at least .80) to conduct the analyses of the objectives using logistic regression.

At the time of enrollment into the study, an educational brochure and a letter will be sent to all potential participants advising them that they may not be up to date in colon cancer screening and that they will be receiving a free FIT test in the mail in a couple weeks. The letter will advise them that they will be participating in a study that Renown is doing to improve the ability to diagnose early colon cancer and that they will be contacted by Renown with their results and also any additional recommendations if the FIT is positive. If they have questions or do not want to participate, there is a number for potential participants to call for more information or to opt out. Patients that choose not to participate in the study who would still like to complete the FIT screening kit, will be informed that they will be responsible to pay for the FIT test (about $25) following Renown's standard operating procedures.

2 weeks after the initial letter, all newly enrolled patients will receive a mailing including a FIT test, an educational brochure, instructions on how to collect the FIT test and a Thank You letter for participating.

An initial automated telephone message will be left for each patient at the time of the mailing reminding them to submit their stool FIT. At 2 and 3 weeks after the FIT mailing all patients medical records will be reviewed and those who have not yet returned their stool FIT will receive an automated telephone call reminder to mail in their stool FIT.

At 4 weeks all patients who have not yet returned their stool FIT will be contacted by phone and those that are able to be reached and agree to submit the stool FIT will be mailed a 2nd stool FIT if needed. If the stool FIT is not submitted by 2 months of the mailing, the patient will be listed as not returning a FIT.

All patients who have returned a stool FIT with a negative result will be provided their results by letter.

The patients PCP will be also provided the positive or negative results by letter.

All patients with a positive stool FIT will be randomized into either Usual Care or Choice study groups. The two study groups will be matched by gender, race/ethnicity, Spanish-speakers, and rural/urban location.

Patients in Group 1 (Usual Care) who have a positive result will be contacted by phone by the Nurse Navigator with their results, receive some education about the significance of a + stool FIT relative to colon cancer screening and advised to make an appointment with a PCP or Gastroenterologist to discuss the results and possibly be referred for colonoscopy. If they do not have a PCP they will receive assistance in being referred to one. They will be asked to complete a telephone questionnaire that explores patient demographics (education, race, income, prior colonoscopy etc) in Spanish or English. Patients' EPIC electronic medical records will be monitored to see if they have made an appointment within 2 days of getting their results. If not, they will receive 2 attempted live telephone reminders followed by a certified letter. If a patient is referred to a GI consult, and fails to schedule an appointment within 1 month, GI will notify the patients Renown PCP of the failed appointment.

Patients in Group 1 with a positive result who cannot be reached by phone will receive a certified letter with their results with instructions to contact the Study Navigator to arrange further testing.

Patients in Group 2 (Choice) who have a positive FIT result will be contacted by phone by the Nurse Navigator with their results, receive some education about the significance of a + stool FIT relative to colon cancer screening and given the choice to either schedule an appointment with a PCP or Gastroenterologist to discuss their results, or will receive direct referral to Gastroenterology Consultants for a colonoscopy. They will be asked to complete a telephone questionnaire that explores patient demographics (education, race, income, prior colonoscopy) in Spanish or English. Patients will then receive assistance and monitoring as in that described above for Group 1 depending upon whether they are referred for an office visit/consultation vs. a direct referral for a colonoscopy.

Patients in Group 2 with a positive result who cannot be reached by phone will receive a certified letter with their results with instructions to contact the Study Navigator to arrange further testing.

Patients who are referred directly for a colonoscopy will be contacted by phone by a scheduler at Gastroenterology Consultants and be asked questions to determine the best bowel preparation and sedation for them (conscious sedation with fentanyl and versed vs. propofol, and to insure that the patient has no significant co-morbidities that might require a pre-colonoscopy visit for medical assessment (anticoagulants, severe lung disease, recent MI, bleeding disorder).

Additionally, those that are referred for a direct colonoscopy and fail to schedule or show for their appointment will be referred back to the Renown Nurse Navigator for 2 attempts at a live call then a certified letter.

All patients in group 2 who have not yet had a colonoscopy 6 months after they were initially given their results will again be contacted by phone by a Navigator and again encouraged to have colonoscopy or at minimum to discuss the procedure/FIT results with either their physician or a Gastroenterologist and be offered assistance to schedule those appointments.

Patients in both groups will have 1 year from the date their initial FIT test is mailed to obtain a colonoscopy as recorded in the EPIC EMR.

All patients with a positive stool FIT who have completed the study either by having a colonoscopy or by not having a colonoscopy at the end of the study period will be mailed a questionnaire assessing various quality parameters of the colon cancer screening experience with a stamped self addressed envelope for return and Thank You letter for their participation including a $10 Amazon gift certificate as a token of appreciation for their time. If the questionnaire is not returned within 2 weeks, they will be sent a 2nd questionnaire and reminder letter. After 2 more weeks, if the questionnaire is not returned the research assistant will contact the patient to offer the choice to complete the survey over the telephone.

To accommodate Spanish speaking only patients, all documents mailed to patients will be written both in English and Spanish versions and Spanish translators will be available to speak with patients by phone to respond to questions or to go over the questionnaires.

Other Items A script will be used for any participants who call with questions (see "Script if participant calls").

To protect participant's identity, only de-identified data will be reviewed by the UNR co-investigator (Paul Devereux). The de-identified data will be stored on a password-protected computer in Paul Devereux's locked office. The data will be transferred to Paul Devereux using a password-protected USB flash drive. Data will not contain, names, addresses, dates of birth, or Renown ID numbers.

ELIGIBILITY:
Inclusion Criteria:

* Participants that have not had a colonoscopy with in 10 years, flexible sigmoidoscopy with in 5 years, or a stool for occult blood with in 1 year.

Exclusion Criteria:

* History of colon cancer, inflammatory bowel disease or colon polyps.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13392 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Colonoscopy Completion | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Devereux, PhD, MPH, Study Chair — Univeristy of Nevada, Reno; John Gray, MD, FACG, Principal Investigator — GI Consulatants
Locations (1):
- Renown Regional Medical Center, Reno, Nevada, United States